CLINICAL TRIAL: NCT02795104
Title: Comparative Effectiveness of Interventions to Improve Screening Among Rural Women
Brief Title: Rural Interventions for Screening Effectiveness
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OSU-16108; NCI-2016-00774 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA196243 (NIH)
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Breast, Cervical or Colorectal Cancer Screening Needed
Keywords: RISE
MeSH Terms: interventions — Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (TIDVD) (Experimental): Educational Intervention via DVD: In this arm of the intervention participants watch a tailored interactive DVD program and answer questions posed by the DVD program.
  Interventions: Behavioral: Educational Intervention via DVD
- Arm II (TIDVD, PN) (Experimental): Educational Intervention-DVD & Telephone based Navigation: In this arm of the intervention participants watch a TIDVD and are called by a patient navigator.
  Interventions: Behavioral: Educational Intervention-DVD & Telephone Based Navigation
- Arm III (UC) (Experimental): Educational Intervention via brochure: In this arm of the intervention participants receive brochures that explain and provide information and encouragement for cancer screening.
  Interventions: Behavioral: Educational Intervention via brochure

INTERVENTIONS:
Behavioral: Educational Intervention via brochure — Educational Intervention via brochure:
  In this arm of the educational intervention the participant receives brochures
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm III (UC)
Behavioral: Educational Intervention via DVD — Educational Intervention via DVD: In this arm of the educational intervention the participant receive a tailored interactive DVD to watch
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (TIDVD)
Behavioral: Educational Intervention-DVD & Telephone Based Navigation — Educational Intervention via Telephone-Based Navigation: In this arm of the educational intervention the participant receives a tailored interactive DVD to watch and telephone calls from a patient navigator
  Arms: Arm II (TIDVD, PN)

SUMMARY:
This randomized clinical trial studies how well a tailored interactive digital versatile disc (DVD) with or without patient navigation works in improving screening rates in rural women for breast cancer, cervical cancer or colorectal cancer. A tailored interactive DVD and patient navigation may help rural women to learn more about cancer screening and to better understand the results.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the effectiveness of a tailored and interactive DVD (TIDVD) versus (vs.) TIDVD + telephone-based patient navigation (PN) intervention (TIDVD + PN) vs. usual care (UC), to increase guideline-based cancer screening rates at 12 months post randomization for breast cancer (BC), cervical cancer (CC), and colorectal cancer (CRC) among 1058 women age 50 to 74 living in rural northwest Ohio and northeast Indiana.

II. Compare the cost effectiveness of the TIDVD and the TIDVD + PN intervention vs. UC, for adherence to each screening outcome or combination of screening tests.

OUTLINE: Patients are randomized to 1 of 3 arms.

Arm I: Patients watch a tailored interactive DVD program and answer questions posed by the DVD program.

Arm II: Patients engage in TIDVD and PN.

Arm III: Patients receive brochures that explain and provide encouragement for cancer screening.

After completion of the study, patients are followed up at 2 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Be non-adherent to one or more recommended screenings for BC, CC, or CRC by Medical Record Review (MRR)
* Reside in one of 32 rural counties in Indiana (IN) or Ohio (OH)
* Provide informed consent
* Able to speak/read English
* Have access to a DVD player or computer that can play DVDs

Exclusion Criteria:

* Have a personal or family history of any hereditary/genetic cancer syndrome such as BRCA1 and BRCA2 polymorphisms, hereditary nonpolyposis colon cancer, or familial adenomatous polyposis
* Have a personal history of inflammatory bowel disease (Crohn's disease or colitis), colon polyps, or a history of cancer except non-melanoma skin cancer
* Have a first degree relative with a history of breast or colorectal cancer
* Plan to move outside of the country within the next year
* Reside in a nursing home or other institution
* Are pregnant or intend to become pregnant during the study period

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center; Victoria Champion, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
These data will only be used to characterize/compare the group individual to those who are eligible and agree to participate; with those who are ineligible and will not be shared after the completion of the study with other researchers.

REFERENCES:
- [Derived] Champion VL, Paskett ED, Stump TE, Biederman EB, Vachon E, Katz ML, Rawl SM, Baltic RD, Kettler CD, Seiber EE, Xu WY, Monahan PO. Comparative Effectiveness of 2 Interventions to Increase Breast, Cervical, and Colorectal Cancer Screening Among Women in the Rural US: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e2311004. doi: 10.1001/jamanetworkopen.2023.11004. PMID 37115541
- [Derived] Biederman E, Baltic R, Katz ML, Rawl S, Vachon E, Monahan PO, Stump TE, Kettler C, Carter L, Young G, Xu W, Paskett ED, Champion V. Increasing breast, cervical, and colorectal cancer screening among rural women: Baseline characteristics of a randomized control trial. Contemp Clin Trials. 2022 Dec;123:106986. doi: 10.1016/j.cct.2022.106986. Epub 2022 Oct 31. PMID 36328234
- See also: The James — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I Tailored and Interactive Digital Versatile Disc (DVD) (TIDVD): TIDVD: In this arm of the intervention participants watch a tailored interactive DVD program and answer questions posed by the DVD program.
- Arm II TIDVD and Patient Navigation (PN) (TIDVD, PN): TIDVD,PN: In this arm of the educational intervention the participant receives a tailored interactive DVD to watch and telephone calls from a patient navigator
- Arm III Usual Care (UC): UC: In this arm of the intervention participants receive brochures that explain and provide information and encouragement for cancer screening.
Period: Overall Study
Arm/Group | Arm I Tailored and Interactive Digital Versatile Disc (DVD) (TIDVD) | Arm II TIDVD and Patient Navigation (PN) (TIDVD, PN) | Arm III Usual Care (UC)
Started | 389 | 395 | 201
Completed | 382 | 388 | 193
Not Completed | 7 | 7 | 8
Not completed — Determined to be Ineligible with Exit Data | 7 | 5 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ARM III (UC): Educational Intervention via brochure: In this arm of the intervention participants receive brochures that explain and provide information and encouragement for cancer screening.
  Educational Intervention via brochure: Educational Intervention via brochure:
  In this arm of the educational intervention the participant receives brochures
- Total: Total of all reporting groups
Arm/Group | ARM I (TIDVD) | ARM II (TIDVD, PN) | ARM III (UC) | Total
Number analyzed (Participants) | 382 | 388 | 193 | 963
Age, Customized [Median (Standard Deviation); unit: years] — Population: Nineteen participants (7 TIDVD, 5 TIDVD,PN, 7 UC) who enrolled and participated in the program were determined to be ineligible through additional cancer screening information obtained via exit medical record review. Two participants in the TIDVD,PN Arm withdrew and asked that their data not be used. Exit medical record data was unable to be obtained for one Usual Care participant. These 22 were excluded from analyses.
  years
    Age at consent | 58.2 (6.4) | 58.8 (6.3) | 58.8 (6.3) | 58.6 (6.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 382 | 388 | 193 | 963
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 376 | 375 | 185 | 936
  More than one race | 3 | 6 | 3 | 12
  Unknown or Not Reported | 1 | 3 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Indiana | 159 | 149 | 70 | 378
  United States: Ohio | 223 | 239 | 123 | 585

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Received All Needed Screening and Any Needed Screening Across the Three Randomized Arms
Description: Will be tested initially with pair-wise chi-square tests. Binary logistic regression analysis will be used to compare the two interventions and the UC group on the binary dependent variable (adherence), while adjusting for any potentially confounding covariates. The models will be controlled for any demographic covariate (e.g., age, education) for which the randomized groups differ significantly at baseline using a liberal significance level of 0.20 to achieve conservative adjustment. As a sensitivity analysis, multiple imputation will be used to impute the adherence outcome for participants.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (TIDVD) | Arm II (TIDVD, PN) | Arm III (UC)
Number analyzed (Participants) | 382 | 388 | 193
Participants
  Received All Needed Screenings within 12-months of Enrollment | 57 | 118 | 19
  Received Any Needed Screening within 12-months of Enrollment | 110 | 189 | 48

2. Secondary Outcome: Cost Effectiveness of Each Intervention
Description: Cost-effectiveness analysis (CEA) implies a comparison of whether the cost per unit of outcome in one situation exceeds that in another. Unless the outcome measures are comparable, this is not possible. Will be able to examine outcomes of the interventions and the UC group (participants who up to date with all three cancer screening guidelines at 12 month follow-up). CEA will consist of measuring the incremental cost of achieving the observed incremental outcomes, but not a cost-effectiveness ratio in standard terms.
Time Frame: Up to 12 months
Population: Same as main outcome. All participants included.
Measure: Number; unit: USD ('22) per completed UTD screening
Arm/Group | ARM I (TIDVD) | ARM II (TIDVD, PN) | ARM III (UC)
Number analyzed (Participants) | 382 | 388 | 193
USD ('22) per completed UTD screening | 14,462.64 | 10,638.20 | 0

3. Secondary Outcome: Cost of the Interventions
Description: In the model implemented in this study, the patient navigators spend full time in that activity. Thus, the costs of implementation are straightforward and obtainable. Even though the navigator is full-time, data were collected concerning broad categories of time use through a structured time log so that the cost of specific components (e.g., arranging transportation) can be estimated more accurately. A developed Participant Encounter Form and a Tracking Log of Direct Participant Contacts were used to provide the majority of this information.
Time Frame: Up to 12 months
Population: Same as main outcome. All participants of study.
Measure: Number; unit: US Dollars (2022)
Arm/Group | ARM I (TIDVD) | ARM II (TIDVD, PN) | ARM III (UC)
Number analyzed (Participants) | 382 | 388 | 193
US Dollars (2022) | 326,012.29 | 670,841.46 | 0

ADVERSE EVENTS:
Time Frame: Participants could report any and all issues to the study team from enrollment to study exit (1 year) via mail, email, fax, or phone.
Arm/Group | Arm I Tailored and Interactive Digital Versatile Disc (DVD) (TIDVD) | Arm II TIDVD and Patient Navigation (PN) (TIDVD, PN) | Arm III Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/382 | 0/388 | 0/193
Serious Adverse Events (participants affected / at risk) | 0/382 | 0/388 | 0/193
Other Adverse Events (participants affected / at risk) | 0/382 | 0/388 | 0/193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02795104/Prot_SAP_000.pdf